CLINICAL TRIAL: NCT06285019
Title: Efficacy and Safety of Modified Hepatic Artery Infusion Chemotherapy (TOMOX-HAIC) in Combination With Sintilimab and Bevacizumab Biosimilar for the First-line Treatment of Advanced Hepatocellular Carcinoma: a Prospective, Single-arm, Phase II Clinical Study
Brief Title: Modified TOMOX-HAIC in Combination With Sintilimab and Bevacizumab Biosimilar for First-line Treatment of Advanced Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lu Wang, MD, PhD, Director of Hepatobiliary Surgery, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWK-2023-004
Record Dates: First submitted 2024-02-21; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combination therapy (Experimental): TOMOX-HAIC combined with Sintilimab and bevacizumab biosimilar
  Interventions: Procedure: TOMOX-HAIC; Drug: Sintilimab; Drug: Bevacizumab

INTERVENTIONS:
Procedure: TOMOX-HAIC — Oxaliplatin 85mg/m^2 plus Raltitrexed 3mg/m^2, 21 days for a cycle
Drug: Sintilimab — 200mg, ivgtt, d1, 21 days for a cycle
Drug: Bevacizumab — 7.5mg/kg, ivgtt, d1, 21 days for a cycle

SUMMARY:
This is a single-center, single-arm, phase II clinical study, to explore the efficacy and safety of modified TOMOX-HAIC combined with sintilimab and bevacizumab biosimilar as first line treatment in patients with advanced hepatocellular carcinoma.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most common malignant tumors worldwide.The IMbrave150 study and the Orient-32 study demonstrated that PD-1 in combination with bevacizumab confers better survival outcomes in advanced hepatocellular carcinoma. In addition, HAIC combined with targeted therapy and immunotherapy has shown good safety and encouraging efficacy. Oxaliplatin-based FOLFOX regimen is currently the mainstream HAIC chemotherapy regimen (FOLFOX HAIC) in China.

The results of the previous study confirmed that raltitrexed shows promising antitumor activity and safety in hepatocellular carcinoma. Also, TOMOX-HAIC regimen can significantly shorten the infusion duration and is expected to improve the patient experience, quality of life, and adherence while ensuring the efficacy.

In this clinical trial, patients will receive TOMOX-HAIC combined with Sintilimab and bevacizumab biosimilar. The primary endpoint is overall response rate. The secondary endpoint are disease control rate, time to progression, duration of response, overall survival, and safety

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Males or unpregnant females who age ≥ 18 years, ≤75 years.
* The investigator believes the patient is capable of complying with the study protocol.
* Histologically, cytologically or clinically confirmed advanced hepatocellular carcinoma.
* is not a candidate for radical surgery
* not received previous systemic treatment
* patients must have at least one measurable lesion (RECIST 1.1)
* ECOG PS：0-1, 14 days before enrollment
* Child-Pugh A or Child-Pugh B ≤ 7, 14 days before enrollment

Exclusion Criteria:

* Prior history of other malignant tumors
* Current or prior immunodeficiency disorders or autoimmune diseases
* Subjects have untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk of bleeding
* Subjects who are not available for follow-up or are participating in other clinical trials that have the potential to interfere with this study
* Conditions considered unsuitable for inclusion by researchers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | 24 months
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1. and mRECIST

SECONDARY OUTCOMES:
disease control rate (DCR) | 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 and mRECIST as assessed by investigator
Progression-Free Survival (PFS) | 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) and mRECIST as assessed by investigator
Time to progression (TTP) | 24 months
  the time from randomization until first evidence of disease progression
Duration of response (DOR) | 24 months
  defined as the time from randomization to disease progression or death in patients who achieve complete or partial response
overall survival (OS) | 24 months
  OS is the time from enrollment to death due to any cause.
adverse event (AE) | 24 months
  using the The NCI Common Terminology Criteria for Adverse Events (NCI CTCAE v5.0)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China